CLINICAL TRIAL: NCT05122676
Title: Patient-centered Team-based Primary Care to Treat Opioid Use Disorder, Depression, and Other Conditions
Brief Title: More Individualized Care: Assessment and Recovery Through Engagement
Acronym: MI-CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Indiana University Health (Other); National Institute of Mental Health (NIMH) (NIH); Boston Medical Center (Other); University of New Mexico (Other); University of Washington (Other); Purdue University (Other); Montana State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UF1MH121949 (NIH); 1UF1MH121949-01 (NIH); 4UF1MH121949 (NIH)
Record Dates: First submitted 2021-10-29; First posted 2021-11-17 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Depression; Anxiety; Opioid-Related Disorders; Pain, Chronic
Keywords: Primary health care; Primary care; Primary care nursing; Evidence-based care; Depressive symptoms; Anxiety disorders and symptoms; Mental Health; Mental Health disorder; Opioid use; Opioid misuse; Opioid use disorder; Opioid dependence; Buprenorphine; Substance use disorders; Overdose; Overdose of opiate; Opioid overdose; Motivational Interviewing; Brief psychotherapy
MeSH Terms: conditions — Depression; Anxiety Disorders; Opioid-Related Disorders; Chronic Pain; Psychological Well-Being; Mental Disorders; Substance-Related Disorders; Drug Overdose; Opiate Overdose

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Usual care arm participants are not informed of the study; their secondary data are used for study analyses. Investigators are masked to all individuals in usual care arm and to the safety monitoring reports shared with the Data and Safety Monitoring Board (DSMB); study arms are masked in safety monitoring reports provided to the Data Safety and Monitoring Board unless the DSMB requests that they be unmasked; and statistical analysts conducting main outcomes are blinded to arm by masking and omission of any data in main analytic datasets that would indicate intervention arm (e.g., any measures related to nurse care managers).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI-CARE program (Experimental): Those automatically identified as eligible and randomized to the MI-CARE arm are outreached by a study nurse care manager and offered the 12-month long virtual Collaborative Care program by telephone or video visits. Individuals are free to accept or decline the offer (e.g., stop/restart, not accept right away) during the 12 months after their randomization date.
  Interventions: Behavioral: More Individualized Care: Assessment and Recovery through Engagement (MI-CARE)
- Usual care (No Intervention): Those identified as eligible and randomized to the usual care arm have no contact with the study. All outcome data for both study arms are collected from secondary, electronic sources.

INTERVENTIONS:
Behavioral: More Individualized Care: Assessment and Recovery through Engagement (MI-CARE) — This study evaluates whether offering nurse collaborative care management for 12 months by telephone or video can improve depression-related symptoms, increase access to evidence-based medication treatment for opioid use problems, as well as decreasing adverse health events. Participants randomized to the nurse support arm can work with the nurse at no cost for up to 12 months via phone or video visits.
  The nurse asks questions about stress, mood, worry, pain, sleep, and medication and substance use; participants choose what to focus on. The nurse meets weekly with clinical consultants who may recommend treatment options, tailored to the patient. The participant and their regular provider(s) can discuss the options and decide which to try. The nurse and primary care provider can then help the patient access selected options. The nurse can also offer behavioral activation to help build skills to increase day-to-day positive adaptive experiences and support broader treatment gains.
  Arms: MI-CARE program

SUMMARY:
The MI-CARE trial tests 12 months of telephone-based nurse care management for patients with depressive symptoms who take or have taken opioids at some time. The study tests whether offering nurse support to the patient and their primary care team that addresses these things and related issues can improve patients' health and well-being. Eligible subjects are identified automatically using health system data and randomly assigned 50:50 to either a no-contact usual care arm or to the arm offered the MI-CARE program.

DETAILED DESCRIPTION:
The MI-CARE trial is a randomized encouragement trial that will test whether offering a primary care-based collaborative care (CC) model can increase opioid use disorder (OUD) treatment and improve depression outcomes among patients with:

1. recent electronic health record (EHR) documentation of depressive symptoms, and
2. evidence of OUD documented in the prior year.

The study objective is to evaluate the effectiveness of offering eligible primary care patients the MI-CARE CC program for up to 12 months when compared to usual primary care. Among all eligible primary care patients, MI-CARE and usual primary care will be compared to assess the following outcomes:

* Aim 1: Days of OUD medication treatment (buprenorphine)
* Aim 2: Improvement of depression symptoms.
* Aim 3 (intervention arm only): Examining a) implementation using mixed-methods formative evaluation including reach, adoption, and implementation fidelity, and b) nurse care manager time needed to support the MICARE intervention.

The MI-CARE CC intervention is offered by a nurse care manager (NCM) and delivered by telephone (or video) visits to consenting patients. The intervention is designed to support "whole health" by engaging patients in medication treatment for OUD and depression, reducing depressive symptoms, and addressing common comorbid conditions that complicate OUD and depression (e.g., anxiety, pain, sleep, and other mental health and substance use disorders).

The Collaborative Care Model was originally designed to improve mental health outcomes in primary care and includes 5 essential elements. The CC intervention tested in the MI-CARE trial will include each of these elements: population-based care, patient-centered team care, evidence-based care, measurement-based treatment to target, and accountable care.

The MI-CARE program begins with NCM care focused on PCP and patient engagement:

* Care team engagement - In addition to engaging the patient, the engagement process is designed to build the relationship between the NCM and the primary care team. Prior to a patient's first outreach call, the NCM informs the PCP that their patient was selected for the CC program and offers to have an initial brief (optional) call about the program with the care team. The NCM may also reach out to engage with specialty mental health providers who are working closely with the patient. If the patient does not have an established PCP, the NCM will offer to work with the patient to establish a PCP within the healthcare system. Additionally, each site's collaborative care consultants will message PCPs in their health plan when a given PCP's patient consents to participate in the MICARE intervention. These messages are to inform the PCP of the support the CC consultants provide each NCM in the management of consented patients to the intervention (including that the CC consultant's role may include various recommendations regarding patient care).
* Patient engagement - This begins with a short series of "engagement" sessions to develop a relationship with the patient. Engagement sessions focus on eliciting a patient's health narrative, including current symptoms, and exploring the patient's (general) health goals, priorities, and preferences. Prior to the first engagement call the NCM reviews the patient's chart to obtain current treatment(s) for depression, OUD and related conditions. The NCM will build rapport by learning about patients' lives, how they are impacted by their health, eliciting the patients' thoughts on symptoms reported, and exploring how the program might help them. Motivational interviewing and shared decision-making techniques are used to elicit patient goals and priorities.

Beginning with engagement and throughout the follow up period, the NCM will use common elements of two evidence-based core behavioral approaches:

* Motivational interviewing (MI) skills to elicit ambivalence and move patients toward wanting to improve OUD, depression or other related conditions; and
* Behavioral activation (BA) to help participants build skills to increase positive adaptive experiences in their day-to-day lives and support broader treatment gains.

ELIGIBILITY:
INCLUSION CRITERIA

Eligible patients must meet all 4 criteria:

1. ≥1 in person or virtual encounter in a primary care setting in the 365 days prior to the data extraction date (pull date);
2. Age ≥18 years at the pull date;
3. ≥1 PHQ-9 depression screening score of ≥10 within the 7 days prior to the pull date.
4. Evidence of potential OUD in the 365 days prior to and including the date of the qualifying PHQ-9 score. Any 1 of the following qualifies as evidence of potential OUD:

   1. ≥1 active OUD ICD-10 diagnosis code in any setting except labs;
   2. ≥1 prescription (orders or dispensed) for buprenorphine (oral formulations indicated for OUD, extended release injectable, and implant);
   3. ≥1 procedure code for buprenorphine (oral formulations indicated for OUD, extended release injectable, and implant);
   4. ≥1 ICD-10 codes for opioid overdose;
   5. ≥1 OUD ICD-10 code, including remission, and prescription (orders or dispensed) or procedure code for injectable naltrexone.

EXCLUSION CRITERIA

Patients are ineligible who meet any of the criteria below:

1. The only indication of OUD or only PHQ available to determine eligibility came from data protected under 42 CFR Part 2;
2. The patient has already been randomized to the trial or was outreached in the pilot study (including outreach to the primary care provider only);
3. English interpreter required (per health system records).
4. Any one of the following conditions in the 2 years prior to and including the date of the qualifying PHQ:

   1. Alzheimer's disease or dementia diagnosis, or medication to treat Alzheimer's or dementia.
   2. Severe cognitive limitations.
5. Current active treatment for cancer with chemotherapy or radiation therapy in the past 3 months (not including non-melanoma skin cancers).
6. Previously requested to not participate in research studies at the health system;
7. Documentation of hospice care in the 2 years prior to and including the date of the qualifying PHQ score;
8. Patient is actively being outreached for (or is participating in) depression care management (Kaiser Permanente Washington only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Days of buprenorphine medication treatment for opioid use disorder (OUD) | days 1-365 after randomization
  A continuous measure of days of OUD treatment with buprenorphine in the 365 days after randomization from secondary electronic data sources.

SECONDARY OUTCOMES:
Change in depressive symptoms | 3-13 months after randomization
  Change in depressive symptoms from the study qualifying Patient Health Questionnaire (PHQ) score to follow-up PHQ score documented as part of routine clinical care 3-13. months later from secondary electronic data sources. The 9-item Patient Health Questionnaire (PHQ9) has a minimum score of 0 and a maximum score of 27. the 2-item Patient Health Questionnaire (PHQ2) has a minimum score of 0 and a maximum score of 6. An increasing PHQ score indicates an increase in depressive symptoms.

OTHER OUTCOMES:
Buprenorphine treatment or improved depressive symptoms | 1 day - 13 months after randomization
  Composite measure identifying whether a patient is treated with buprenorphine and/or has documentation of clinically-significant improvement in depressive symptoms from secondary electronic data sources:
  * Treatment with buprenorphine is a binary measure of treatment with buprenorphine formulations for pain or OUD defined as > 90 days of buprenorphine during the 12-month follow up period.
  * Clinically significant improvement in depressive symptoms is a binary measure of documented clinical response of depressive symptoms during follow-up (50% decrease in PHQ9 score or negative PHQ2 screen).
Major acute adverse health events | 12 months after randomization
  A composite of any major adverse event over 12 months of follow-up, which includes: opioid overdose, other drug overdose, suicide attempt or other self-harm, hospitalizations (opioid and non-opioid), or death (from secondary electronic data sources).
Serious opioid related event | 12 months after randomization
  A count of the number of serious opioid-related events over 12 months of follow up; defined as emergency department visits or hospital admissions with a primary OUD or opioid-related diagnosis or an opioid-related overdose (lethal of non-lethal), from secondary electronic data sources.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn DeBar, PhD, Principal Investigator — Kaiser Permanente; Katharine A Bradley, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Indiana University Health, Indianapolis, Indiana
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The MI-CARE trial will involve analysis of a large amount of detailed proprietary secondary electronic health plan data from the Kaiser Permanente Washington and Indiana University Health systems, and state-wide datasets, e.g., prescription monitoring programs (PMPs). We will seek to obtain data use agreements that allow us to share all de-identified data. However, if that is not possible, we will share those de-identified data for which we do have permission to share.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Access Criteria: Although our trial had planned to publicly share data with the NIMH data archive (NDA), they determined on February 24, 2022 that they would remove our grant from NDA data sharing because the subjects in this trial do not have signed consent forms.

REFERENCES:
- [Derived] DeBar LL, Bushey MA, Kroenke K, Bobb JF, Schoenbaum M, Thompson EE, Justice M, Zatzick D, Hamilton LK, McMullen CK, Hallgren KA, Benes LL, Forman DP, Caldeiro RM, Brown RP, Campbell NL, Anderson ML, Son S, Haggstrom DA, Whiteside L, Schleyer TKL, Bradley KA. A patient-centered nurse-supported primary care-based collaborative care program to treat opioid use disorder and depression: Design and protocol for the MI-CARE randomized controlled trial. Contemp Clin Trials. 2023 Apr;127:107124. doi: 10.1016/j.cct.2023.107124. Epub 2023 Feb 18. PMID 36804450

DOCUMENTS (1):
  • Study Protocol (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT05122676/Prot_003.pdf